CLINICAL TRIAL: NCT06195800
Title: Identifying Immune Biomarkers of Disease and Disease Control in Autoimmune Neurological Disease Using Autologous Haematopoietic Stem Cell Transplantation
Brief Title: Biomarkers of aHSCT
Acronym: BIO-MS
Status: Recruiting | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Sheffield Hospitals Charity (Unknown); Nottingham Trent University (Other); University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH22343
Record Dates: First submitted 2023-10-13; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: multiple sclerosis; aHSCT; Autologous haematopoetic stem cell transplantation
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Stem cells Stool/microbiome Mucosal Cerebrospinal fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated with aHSCT: Patients with aggressive disease treated with autologous haematopoetic stem cell transplantation.
- Patients treated with disease modifying treatment: Patients with aggressive disease treated with high efficacy disease modifying treatment

SUMMARY:
The underlying disease mechanisms which occur in patients with immune mediation neurological diseases, such as Multiple Sclerosis (MS), are incompletely understood. For such patients, autologous haematopoietic stem cell transplantation (aHSCT) has been increasingly used as a highly successful one-off treatment for some patients. This treatment aims to delete the faulty immune system with a course of chemotherapy and then 'reboot' the immune system using a patients' own stem cells (a cell with the unique ability of being a building block to create many different cells in the body) to stop further damage. Over the last 20 years more than 1800 patients with MS have been treated in Europe with high levels of success. It may be more successful than disease modifying treatment but unfortunately, a small portion of people do not respond to this treatment optimally and continue to accumulate disability. There is a risk of side effects, restricted largely to the time of treatment, which necessitates the need to ensure appropriate patients are treated. Whilst aHSCT is a very effective therapy, it is still in its early phase of development, is not in widespread use, and there is incomplete knowledge regarding how it works and importantly, why it does not work in some patients, and how to monitor response to treatment.

Unfortunately, there is no way of detecting which patients will, and will not, benefit from the different treatments available or a way of monitoring the immune system to ensure further treatment is provided before irreversible damage occurs.

This study will investigate the immune system which is found in the fluid surrounding the brain and spinal cord, blood and stool of patients undergoing aHSCT and compare it to those receiving disease modifying treatment. This study will therefore further the understanding of biomarkers of aHSCT to develop an awareness of how it can be refined, may improve monitoring of patients following treatment and permit the development of markers which can predict potential treatment success or failure before patients are exposed to the risks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of a immune mediated neurological disease according to disease specific criteria (active treatment arm) or diagnosis of relapsing remitting multiple sclerosis (control arm).
2. Treatment with autologous haematopoetic stem cell transplantation (active treatment arm) or high efficacy disease modifying treatment (control arm).
3. Willing to provide biological samples for analysis and undergo clinical assessments for the duration of follow up.
4. Able to understand English and provide informed consent.

Exclusion Criteria:

1. Inability to provide informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients who are attending the Sheffield (UK) transplant clinic for neurological disease.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2026-08-09 (Estimated); Study Completion 2026-08-09 (Estimated)

PRIMARY OUTCOMES:
Quantitatively and qualitatively characterise the immune profile of the stem cells, blood, cerebrospinal fluid (CSF) and the microbiome pre and post treatment. | 24 months
  Phenotype profiling of stem cells, cells in blood and CSF using multi-parameter flow cytometry.
  Profile the gut microbiome using 16S rRNA sequencing and flow cytometric analysis.
Perform single cell RNA sequencing (scRNA-Seq) on paired CSF and blood pre and post treatment. | 24 months
  Profiling of T cell receptor and B cell receptor repertoire diversity and clonality

SECONDARY OUTCOMES:
Characterisation of the regeneration of mucosal cell immunity and the reconstitution of pathogen specific immunity following aHSCT by scRNA-Seq on nasopharyngeal swabs and mucosal strips. | 24 months
  Assess immune response in treated patients post vaccination.
Evaluate immunological disease response and the duration of response to aHSCT according to expanded disability status scale score (EDSS) | 24 months
  EDSS to be observed longitudinally following treatment.
Evaluate immunological disease response and the duration of response to aHSCT according to low contrast visual acuity (LCLA) | 24 months
  LCLA to be observed longitudinally following treatment.
Evaluate immunological disease response and the duration of response to aHSCT according to multiple sclerosis functional composite score (MSFC) | 24 months
  MSFC to be observed longitudinally following treatment.
Evaluate immunological disease response and the duration of response to aHSCT according to short form 36 (SF-36) | 24 months
  SF-36 to be observed longitudinally following treatment.
Evaluate immunological disease response and the duration of response to aHSCT according to symbol digit modality test (SDMT) | 24 months
  SDMT to be observed longitudinally following treatment.
Evaluate immunological disease response and the duration of response to aHSCT according to Karnofsky performance status | 24 months
  Karnofsky performance status to be observed longitudinally following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Brittain, MBBS, MRCP, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust and The University of Sheffield
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided